CLINICAL TRIAL: NCT00878202
Title: Impact of Clinical Follow-up and Therapeutic Education by Telemedicine in Chronic Heart Failure: a Randomized Multicenter Study.
Brief Title: Therapeutic Education by Telemedicine in Chronic Heart Failure
Acronym: SEDIC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B80909-60
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Optimal medical treatment of Heart failure and therapeutic education
- Telemedicine (Experimental): Optimal medical treatment of heart failure disease and therapeutic education
  Interventions: Device: SCAD information system

INTERVENTIONS:
Device: SCAD information system — Clinical follow-up and continuation of therapeutic education by telemedicine during 3 months
  Arms: Telemedicine

SUMMARY:
The purpose of the SEDIC study is to test a home based heart failure patient clinical follow-up and therapeutic education using telemedicine. This educational follow-up is based on an interactive information system (SCAD) including a touch screen personal computer for heart failure patient at home. An interactive algorithm has been developed to allow a self management teaching to the patient.Furthermore, a specialized nurse provide a clinical data follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 65 years old hospitalized for acute heart failure
* Left ventricle systolic Dysfunction with ejection fraction < 45 %, documented in the previous 6 months
* And at least one of the following criteria:

BNP before discharge from hospital > 350 pg/ml / EF < 35 % / Hospitalization for acute heart failure informed in the previous 6 months

Exclusion Criteria:

* NYHA 4 at hospital discharge
* Planned cardiac surgery or coronary revascularization
* Hospitalization for ST-elevation acute coronary syndrome
* Depressive syndrome with score > 20 at geriatric depression scale
* Therapeutic education impossible
* Technical problems with the device
* Limited autonomy for device use
* Patient not living in Basse-Normandie
* Ongoing participation in another clinical trial

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of hospitalization days for heart failure | 12 months

SECONDARY OUTCOMES:
Cardiovascular mortality | 12 months
Total mortality | 12 months
Rate of hospitalization for heart failure | 12 months
Median of time up to mortality or hospitalization for heart failure | 12 months
Number of medical consultation | 12 months
Pharmaco-economic analysis | 12 months
Disease knowledge questionnaire | 12 months
Quality of life questionnaire ( Minnesota) | 12 months
BNP | 12 months
Six minutes walk test | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Sabatier, MD, Principal Investigator — University Hospital, Caen; Annette Belin, MD, Principal Investigator — University Hospital, Caen
Locations (6):
- France (6):
  - Alençon-Mamers Hospital, Alençon
  - Caen University Hospital, Caen
  - Cherbourg Hospital, Cherbourg
  - Flers Hospital, Flers
  - Lisieux Hospital, Lisieux
  - Saint-Lo Hospital, Saint-Lô